CLINICAL TRIAL: NCT05208047
Title: A Phase 3 Randomized, Open-Label, Multicenter Clinical Study of CGT9486+Sunitinib vs. Sunitinib in Subjects With Locally Advanced, Unresectable, or Metastatic Gastrointestinal Stromal Tumors
Brief Title: (Peak) A Phase 3 Randomized Trial of CGT9486+Sunitinib vs. Sunitinib in Subjects With Gastrointestinal Stromal Tumors
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cogent Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGT9486-21-301
Record Dates: First submitted 2021-12-23; First posted 2022-01-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Advanced Gastrointestinal Stromal Tumors; Metastatic Cancer
Keywords: Sunitinib; Solid Tumors; Gastrointestinal Stromal Tumors; Gastrointestinal; KIT; Kinase Inhibitors; Growth Inhibitors; CGT9486; Unresectable; Metastatic; GIST; Bezuclastinib; PLX9486; Midazolam; Drug-drug interaction
MeSH Terms: conditions — Neoplasm Metastasis; Gastrointestinal Stromal Tumors | interventions — Sunitinib; Midazolam

STUDY DESIGN:
Intervention Model Description: This is a multi-part study: Part 1a is a single-arm design, Part 1b is a two-arm parallel design drug-drug interaction evaluation in the first treatment cycle and single-arm design in subsequent treatment cycles, and Part 2 is a randomized two-arm parallel comparator study. The DDI substudy is a single-arm, fixed-sequence, crossover design to investigate the potential for CGT9486 to be a CYP3A4 inducer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1a (Experimental): CGT9486 plus sunitinib 37.5 mg QD
  Interventions: Drug: CGT9486 plus sunitinib
- Part 2 - Experimental Group (Experimental): CGT9486 plus sunitinib 37.5 mg QD
  Interventions: Drug: CGT9486 plus sunitinib
- Part 2 - Control Group (Active Comparator): sunitinib 37.5 mg QD
  Interventions: Drug: Sunitinib
- Part 1b - DDI Cohort 1 (Experimental): CGT9486 plus sunitinib 37.5 mg QD
  Interventions: Drug: CGT9486
- Part 1b - DDI Cohort 2 (Experimental): sunitinib 37.5 mg QD plus CGT9486
  Interventions: Drug: Sunitinib
- DDI Substudy (Midazolam) (Experimental): Midazolam, CGT9486, sunitinib
  Interventions: Drug: Midazolam; Drug: CGT9486 plus sunitinib

INTERVENTIONS:
Drug: CGT9486 plus sunitinib — Participants will receive both CGT9486 and sunitinib orally until study stopping rules are met.
  Arms: Part 1a; Part 2 - Experimental Group
Drug: CGT9486 — Participants will receive CGT9486 until steady state then both CGT9486 and sunitinib orally until study stopping rules are met.
  Arms: Part 1b - DDI Cohort 1
Drug: Sunitinib — Participants will receive sunitinib until steady state then both sunitinib and CGT9486 orally until study stopping rules are met.
  Other Names: sunitinib - Part 1b
  Arms: Part 1b - DDI Cohort 2
Drug: Sunitinib — Participants will receive sunitinib orally until study stopping rules are met.
  Other Names: sunitinib - Part 2
  Arms: Part 2 - Control Group
Drug: Midazolam — Participants will receive a single-dose of midazolam on Day 1 and Day 16
  Arms: DDI Substudy (Midazolam)
Drug: CGT9486 plus sunitinib — Patients will receive CGT9486 orally starting on Day 2 and sunitinib starting on Day 16 until study stopping rules are met.
  Arms: DDI Substudy (Midazolam)

SUMMARY:
This is a Phase 3, open-label, international, multicenter study of CGT9486 in combination with sunitinib. This is a multi-part study that will enroll approximately 442 patients. Part 1 consists of two evaluations: 1) confirming the dose of an updated formulation of CGT9486 to be used in subsequent parts in approximately 20 patients who have received at least one prior line of therapy for GIST and 2) evaluating the potential for drug-drug interactions between CGT9486 and sunitinib in approximately 18 patients who have received at least two prior tyrosine kinase inhibitors (TKIs) for GISTs. The second part of the study will enroll approximately 388 patients who are intolerant to, or who failed prior treatment with imatinib only and will compare the efficacy of CGT9486 plus sunitinib to sunitinib alone with patients being randomized in a 1:1 manner. Additionally, a drug-drug interactions substudy will investigate the potential for CGT9486 to be a CYP3A4 inducer in approximately 16 patients who have received at least one prior line of therapy for GIST.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed locally advanced, metastatic, and/or unresectable GIST. Molecular pathology report must be available for Part 2; if molecular pathology report is unavailable or inadequate, an archival or fresh tumor tissue sample will be required to evaluate mutational status prior to randomization.
2. Documented disease progression on or intolerance to imatinib
3. Subjects must have received the following treatment:

   DDI Substudy/Part 1a: Treatment with ≥1 prior lines of therapy for GIST Part 1b: Treatment with ≥2 prior TKI for GISTs Part 2: Prior treatment with imatinib only
4. Have at least 1 measurable lesion according to mRECIST v1.1 (Part1a, Part 1b, Part 2)
5. ECOG - 0 to 2
6. Have clinically acceptable local laboratory screening results (clinical chemistry and hematology) within certain limits

Key Exclusion Criteria:

1. Known PDGFR driving mutations or known succinate dehydrogenase deficiency
2. Clinically significant cardiac disease
3. Major surgeries (eg, abdominal laparotomy) within 4 weeks of the first dose of study drug
4. Gastrointestinal abnormalities including, but not limited to, significant nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude adequate absorption
5. Any active bleeding excluding hemorrhoidal or gum bleeding
6. Seropositive for HIV 1 or 2, or positive for hepatitis B surface antigen or hepatitis C virus (HCV) antibody.
7. Active, uncontrolled, systemic bacterial, fungal, or viral infections at Screening
8. Received strong CYP3A4 inhibitors or inducers
9. Received sunitinib within 3 weeks (Part 1a, Part 1b, DDI Substudy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Part 1a - pharmacokinetics - Cmax | 16 days
  Maximum plasma concentration (Cmax)
Part 1a - pharmacokinetics - AUC | 16 days
  Area under the plasma concentration-time curve (AUC)
Part 1b - pharmacokinetics - Cmax | 14 days
  Maximum plasma concentration (Cmax)
Part 1b - pharmacokinetics - AUC | 14 days
  Area under the plasma concentration-time curve (AUC)
Part 1b - pharmacokinetics - Tmax | 14 days
  Time to maximum observed plasma concentration (Tmax)
Part 2 - Progression Free Survival (PFS) | Approximately 48 months
  Time from first dose to documented disease progression or death due to any cause, whichever occurs first
DDI Substudy - pharmacokinetics - AUC | 16 days
  Area under the plasma concentration-time curve (AUC)
DDI Substudy - pharmacokinetics - Cmax | 14 days
  Maximum plasma concentration (Cmax)

SECONDARY OUTCOMES:
All Study Parts - observing the safety of each treatment regimen. | Approximately 48 months
  Incidence and severity of Adverse Events from first dose of study drug
All Study Parts - observing the safety of each treatment regimen. | Approximately 48 months
  Incidence and severity of Serious Adverse Events from first dose of study drug
All Study Parts - observing the safety of each treatment regimen. | Approximately 48 months
  Incidence of Adverse Events leading to dose modifications from first dose of study drug
All Study Parts - observing the safety of each treatment regimen. | Approximately 48 months
  Change from baseline in laboratory results
Part 1a, Part 1b, Part 2 - Overall Survival (OS) | Approximately 48 months
  Time from first dose to death due to any cause
Part 1a, Part 1b, Part 2 - Objective Response Rate (ORR) | Approximately 48 months
  Percentage of subjects who achieved documented complete response (CR) + confirmed partial response (PR) based on modified Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Part 1a, Part 1b, Part 2 - Disease Control Rate (DCR) | Approximately 48 months
  Percentage of subjects who achieved CR + PR + stable disease (SD) at 16 weeks
Part 1a, Part 1b. Part 2 - Time to response (TTR) | Approximately 48 months
  Time from first dose to first documented response based on modified Response Evaluation Criteria in Solid Tumors Version 1.1
Part 1a, Part 1b, Part 2 - Duration of Response (DOR) | Approximately 48 months
  Time from first response (CR or PR) to the date of progression or death from any cause, whichever occurs first
Part 2 Only - European Organisation for Research and Treatment of Cancer Quality of Life (EORTC-QLQ-30) | Approximately 48 months
  Change in individual scores in patients with locally advanced, unresectable, or metastatic GIST treated with CGT9486 in combination with sunitinib compared with patients treated with sunitinib monotherapy. The scale comprises 30 questions, 24 of which are aggregated into 9 multi-item scales, to include 5 functioning scales (physical, role, cognitive, emotional and social), 3 symptom scales (fatigue, pain and nausea/vomiting) and 1 global health status scale. The remaining 6 single-item scales assess symptoms (dyspnea, appetite loss, sleep disturbance, constipation, diarrhea and the financial impact). All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning, while higher scores on the symptom and single-item scales indicate a higher level of symptoms.

CONTACTS AND LOCATIONS:
Locations (110):
- United States (32):
  - Mayo Clinic, Scottsdale, Arizona
  - University of Arizona- Cancer Center, Tucson, Arizona
  - City of Hope, Duarte, California
  - University of California, Los Angeles (UCLA), Los Angeles, California
  - University of California, San Diego (UCSD), San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Denver, Denver, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Durham, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin - Carbone Cancer Center, Madison, Wisconsin
- Argentina (2):
  - Instituto Alexander Fleming, Buenos Aires
  - Instituto Oncologico de Cordoba (IONC), Córdoba
- Australia (2):
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Bankstown-Lidcombe Hospital, Bankstown
- Brazil (3):
  - Hospital das Clinicas da Universidade Estadual de Campinas (UNICAMP), Campinas
  - lnstituto Nacional de Cancer - INCA, Rio de Janeiro
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, São Paulo
- Canada (4):
  - Alberta Health Services Cross Cancer Institute, Edmonton, Alberta
  - Princess Margaret Hospital, Toronto, Ontario
  - Tom Baker Cancer Center, Calgary
  - Universite de Montreal - Hopital Maisonneuve-Rosemont (HMR), Montreal
- Chile (2):
  - Instituto Oncologico FALP, Santiago
  - Centro de Oncologia de Precision, Universidad Mayor, Santiago
- Czechia (2):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Olomouc - Oncology clinic, Olomouc
- Aarhus University Hospital, Aarhus, Denmark
- France (8):
  - Institut Bergonie, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - AP-HM - Hôpital de la Timone, Marseille
  - Centre Eugene Marquis, Rennes
  - ICO St-Herblain, Saint-Herblain
  - CHU de Toulouse - Hospital Rangueil, Toulouse
  - Gustave Roussy, Villejuif
- Germany (6):
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Helios Klinikum Berlin-Buch, Berlin
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover- Urology Oncology, Hanover
  - Universitaetsmedizin Mannheim, Mannheim
- Hong Kong (2):
  - Hong Kong United Oncology Centre, Jordon
  - Prince of Wales Hospital, Shatin
- Debreceni Egyetem, Klinikai Központ, Onkológiai Klinika, Debrecen, Hungary
- Italy (11):
  - Centro Riferimento Oncologico - Aviano, Aviano
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna - Policlinico di Sant'Orsola, Bologna
  - ASST degli Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori", Meldola
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Policlinico Universitario Campus Bio-Medico, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Ospedaliera Universitaria Integrata Verona-Ospedale Borgo Trento, Verona
- I Can Oncology Center SA De CV, Monterrey, Mexico
- Netherlands (4):
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek Ziekenhuis (NKI-AVL), Amsterdam
  - UMC Groningen, Groningen
  - Stichting Radboud Universitair Medisch Centrum, Nijmegen
  - Erasmus MC, Rotterdam
- Norway (2):
  - Haukeland University Hospital - Bergen, Bergen
  - Oslo University Hospital, Oslo
- Poland (3):
  - Szpital Specjalistyczny w Brzozowie, Brzozów
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Oddzial w Gliwicach, Oddzial Chemioterapii Dziennej, Gliwice
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Klinika Nowotworow Tkanek Miekkich, Kosci i Czerniakow, Warsaw
- South Korea (4):
  - Seoul National University Hosptial, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (8):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Institut Catala d'Oncologia - L'Hospitalet, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
- Sweden (2):
  - Skane University Hospital Lund, Lund
  - Karolinska University Hospital, Solna
- Taiwan (5):
  - Chang Gung Memorial Hospital - Kaohsiung Branch, Kaohsiung City
  - National Taiwan University Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taipei Veterans General Hospital (VGHTP), Taipei
  - Chang Gung Memorial Hospital - Linkou Branch (CGMHLK), Taoyuan District
- United Kingdom (5):
  - Cambridge Addenbrooke's Hospital, Cambridge
  - University College London Hospital, London
  - Royal Marsden Hospital - Surrey, London
  - The Christie NHS Foundation Trust, Manchester
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: No